CLINICAL TRIAL: NCT05256251
Title: Westlake Longevity Cohort
Acronym: We-Longevity
Status: Recruiting | Type: Observational
Sponsor: Westlake University (Other)
Responsible Party: Sponsor
Other Study IDs: 20211015ZJS001
Record Dates: First submitted 2021-11-15; First posted 2022-02-25 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-03

CONDITIONS: Aging
Keywords: Gut microbiome; Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Westlake Longevity Cohort (We-Longevity) is a prospective cohort study among centenarians, nonagenarians and senior citizens living in Lishui, China. The primary aim of this cohort is to characterize the multi-omics molecular characteristics of healthy longevity and their dynamic trajectories. The second aim is to culture the gut microbiota of these elderly people through culturomics. The third aim of We-Longevity is to investigate the association of dietary and lifestyle with the multi-omics molecular characteristics of healthy longevity, and to facilitate the development of personalized nutritional/lifestyle recommendation for the public.

DETAILED DESCRIPTION:
Aging is a major risk factor for most fatal diseases, such as Alzheimer's disease, type 2 diabetes, cardiovascular disease, and cancer. Global population aging is becoming increasingly serious, and this trend is mainly driving the annual increase in the prevalence of aging-related diseases. Healthy longevity is influenced by a variety of factors, such as diet structure, lifestyle, ecological environment, gut microbiome, and genetics. At present, research on healthy longevity is mainly focused on Drosophila, nematodes, and mouse models, but few studies have targeted longevity populations. Centenarians and nonagenarians are the best populations to study healthy longevity. However, the multi-omics molecular characteristics and regulatory mechanisms of healthy longevity in humans are still unclear. Therefore, the We-Longevity design includes centenarians, nonagenarians, and senior citizens. We will determine the fecal/serum metabolome, culturable gut microbiome characteristics, gut microbiome, serum proteome, and genome, together with diet, lifestyle, and disease information.

ELIGIBILITY:
Inclusion Criteria:

* Participants live in Lishui, China.
* Participants intend to remain in Lishui for ≥3 years.

Exclusion Criteria:

* Participants with infectious diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the participants should be Chinese residents, regardless of the ethics.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-11-14 (Estimated); Study Completion 2031-11-14 (Estimated)

PRIMARY OUTCOMES:
Physical frailty | 36 months
  Physical frailty will be evaluated by using Fried's criteria.
Gut microbiome | 36 months
  Fecal microbiome will be analyzed by 16S/ITS rRNA gene sequencing and metagenome sequencing. Furthermore, fecal microbiota will be cultured, picked and identified.

SECONDARY OUTCOMES:
Cognitive function | 36 months
  Cognitive function will be evaluated by using Mini-Mental State Examination (MMSE).
Blood biochemical parameters | 36 months
  Blood biochemical parameters (e.g., glucose and lipids) will be analyzed by an automated biochemical analyzer.
Metabolomics profiling | 36 months
  Blood and fecal metabolomics will be analyzed by LC-MS/MS.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Sheng Zheng, PhD, Principal Investigator — Westlake University
Locations (1):
- Lishui Yikang Hospital, Lishui, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided